CLINICAL TRIAL: NCT04438096
Title: A Randomized, Double-Blind, Parallel Group, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of CVI-LM001 in Patients With Hypercholesterolemia
Brief Title: Safety and Efficacy of CVI-LM001 in Patients With Hypercholesterolemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CVI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVI-LM001-Ⅱ-01
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 100 mg (Experimental)
  Interventions: Drug: 100 mg
- 200 mg (Experimental)
  Interventions: Drug: 200 mg
- 300 mg (Experimental)
  Interventions: Drug: 300 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 100 mg — One 100 mg pill and two placebo pills (QD) will be orally administered for 12 weeks
  Arms: 100 mg
Drug: 200 mg — Two 100 mg pills and one placebo pill (QD) will be orally administered for 12 weeks
  Arms: 200 mg
Drug: 300 mg — Three 100 mg pills (QD) will be orally administered for 12 weeks
  Arms: 300 mg
Drug: Placebo — Three placebo pills (QD) will be orally administered for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if CVI-LM001 is effective and safe versus placebo in drug-naive subjects with elevated LDL cholesterol. There will be 4 groups receiving 100mg, 200mg, 300 mg and placebo treatment for 12 weeks respectively.

DETAILED DESCRIPTION:
This study is a phase II study in subjects with elevated LDL cholesterol. As designed, the study will start with a 4-week, single-blind, placebo run-in period based on diet and exercise interventions for screening eligible subjects. After run-in, eligibility is confirmed with required laboratory tests at Day -1 prior to randomization. The eligible subjects are randomly assigned to CVI-LM001 100 mg, 200 mg, 300mg QD group or placebo QD group with ratio 1:1:1:1 to receive a 12-week double-blind treatment. After 12-week treatment, all investigational compound and placebo should be discontinued, followed by 4 week for safety evaluation.

ELIGIBILITY:
Key Inclusion Criteria:

* 1. Aged 18-70 years, inclusive
* 2. Men and nonpregnant, nonlactating women
* 3. Hypercholesterolemic subjects with LDL-C level between 3.36mmol/L~4.88mmol/L at screening, inclusive

Exclusion Criteria:

* 1. Fasting TG ≥3.99 mmol/L before randomization
* 2. History of significant cardiovascular , renal, pulmonary and liver diseases
* 3. History of diabetes
* 4. ALT or AST>1.5XULN at screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline to Week 12 in Low-density Lipoprotein Cholesterol (LDL-C) | 12 weeks
  The percent change of LDL-C from baseline by comparing CVI-LM001 arms with placebo after 12 weeks of treatment
From Baseline to Week 12 in Number of Participants with Treatment-Emergent Adverse Events | 12 weeks
  Comparison treatment-emergent adverse events of LM001 arms with placebo arm after 12 weeks of treatment

SECONDARY OUTCOMES:
Percent Change From Baseline to Week 12 in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) | 12 weeks
  The percent change of Non-HDL-C from baseline by comparing CVI-LM001 arms with placebo after 12 weeks of treatment
Percent Change From Baseline to Week 12 in Total Cholesterol (TC) | 12 weeks
  The percent change of TC from baseline by comparing CVI-LM001 arms with placebo after 12 weeks of treatment
Percent Change From Baseline to Week 12 in Apolipoprotein B (ApoB) | 12 weeks
  The percent change of ApoB from baseline by comparing CVI-LM001 arms with placebo after 12 weeks of treatment
Percent Change From Baseline to Week 12 in Triglyceride (TG) | 12 weeks
  The percent change of TG from baseline by comparing CVI-LM001 arms with placebo after 12 weeks of treatment
Percent Change From Baseline to Week 12 in High-sensitivity C-reactive Protein (hsCRP) | 12 weeks
  The percent change of hsCRP from baseline by comparing CVI-LM001 arms with placebo after 12 weeks of treatment
Percent Change From Baseline to Week 12 in Lipoprotein（ a）(Lp(a)) | 12 weeks
  The percent change of Lp(a) from baseline by comparing CVI-LM001 arms with placebo after 12 weeks of treatment
Percent Change From Baseline to Week 12 in Proprotein Convertase Subtilisin/Kexin Type 9(PCSK9) | 12 weeks
  The percent change of PCSK9 from baseline by comparing CVI-LM001 arms with placebo after 12 weeks of treatment
Percent Change From Baseline to Week 12 in Apolipoprotein A1 (Apo A1) | 12 weeks
  The percent change of Apo A1 from baseline by comparing CVI-LM001 arms with placebo after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Que Liu, MDPhD, Study Chair — CVI Pharmaceuticals
Locations (1):
- The second affiliated hospital of zhejiang University school of medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
lipid panel including LDL as well as safety data
Supporting Information: Study Protocol
Time Frame: July, 2021